CLINICAL TRIAL: NCT02144857
Title: Effects of Treatment With Biological Agents on Endothelial Glycocalyx,Arterial Elastic Properties, Coronary Flow, Myocardial Deformation and Twisting in Psoriasis. Comparative Study With Patients With CAD or Untreated Hypertension.
Brief Title: Effects of Treatment With Biological Agents on Vascular and Cardiac Function in Psoriasis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Athens (Other)
Responsible Party: Principal Investigator, Ignatios Ikonomidis, Assistant Professor in Cardiology, University of Athens
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 213/19-6-12
Record Dates: First submitted 2014-05-12; First posted 2014-05-22 (Estimated); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Etanercept; Ustekinumab; Cyclosporine; secukinumab; apremilast

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Anti-TNFa regimen (Active Comparator): Etanercept 50 mg
  Interventions: Drug: etanercept
- Anti IL12/23 regimen (Active Comparator): ustekinumab 45 mg
  Interventions: Drug: ustekinumab
- Cyclosporine regimen (Active Comparator): Cyclosporine 2.5-3 mg/kg
  Interventions: Drug: cyclosporine
- anti-interleukin 17 A regimen (Active Comparator): secukinumab 300 mg
  Interventions: Drug: Secukinumab
- inhibitor of phosphodiesterase-4 (Active Comparator): apremilast 30mg
  Interventions: Drug: Apremilast

INTERVENTIONS:
Drug: etanercept — 50 mg
  Other Names: Enbrel
  Arms: Anti-TNFa regimen
Drug: ustekinumab — 45 mg
  Other Names: Stelara
  Arms: Anti IL12/23 regimen
Drug: cyclosporine — Cyclosporine 2.5-3 mg/kgr
  Other Names: Neoral
  Arms: Cyclosporine regimen
Drug: Secukinumab — 300 mg
  Other Names: Cosentyx
  Arms: anti-interleukin 17 A regimen
Drug: Apremilast — 30mg
  Other Names: Otezla
  Arms: inhibitor of phosphodiesterase-4

SUMMARY:
Psoriasis has been associated with an increasing risk for atherosclerosis. The investigators investigated whether surrogate markers of subclinical atherosclerosis, vascular dysfunction and myocardial dysfunction are impaired in patients with psoriasis compared to normal controls ,coronary artery disease patients and untreated hypertension subjects. The investigators also examined the effect of treatment with biological vs no biological agents on vascular and LV function in psoriasis.

DETAILED DESCRIPTION:
The investigators will compare patients with psoriasis with age and sex matched normal controls as well as patients with angiographically documented CAD and patients with untreated hypertension (HYP) used as positive control groups

Patients with psoriasis (PS) will be randomized to receive an anti-tumor necrosis-a (TNF-a) ,an anti- interleukin 12/23 regimen, an interleukin 17A antagonist, apremilast (inhibitor of phosphodiesterase-4) or a cyclosporine regimen.

The anti-TNF-agent, Etanercept will be given at a dose 50mg twice weekly for 12 weeks and after then once weekly.

The anti-IL12/23 regimen, Ustekinumab will be given at a dose 45 mg at the first visit, at 4 weeks and every 12 weeks if body weight is up to 90 kgr. For body weight >90kgr dose will be adjusted accordingly.

The IL-17A antagonist regimen namely secukinumab 300 mg SC at weeks 0, 1, 2, 3, and 4 and 300 mg SC once monthly afterwards Apremilast will be given at a dose of 30mg orally twice daily Cyclosporine will be administered at a dose 2.5-3mg/kgr daily.

At baseline , after 12 weeks and one year of treatment, the investigators will measure:

1. pulse wave velocity (PWVc) augmentation index (AI) central systolic blood pressure (cSBP) (Complior, Alam Medical and Arteriograph,TensioMed)
2. flow-mediated dilation of the brachial artery (FMD)
3. carotid intima-media thickness (IMT) by ultrasonography
4. coronary flow reserve of the LAD (CFR) by Doppler echocardiography
5. E'/A of mitral annular velocities ,LV longitudinal (GLS -%),strain, and strain rate (LongSr-l/s), peak twisting (Tw -deg),peak twisting (Tw-deg/sec)velocity,untwisting at mitral valve opening (unTw) and untwisting (unTw) velocity using speckle tracking echocardiography .
6. Perfused boundary region (PBR)of the sublingual arterial microvessels (ranged from 5-25 microns) using Sideview Darkfield imaging. (Microscan, Glycocheck) .The PBR in microvessels is the cell-poor layer which results from the phase separation between the flowing red blood cells (RBC) and plasma.The PBR includes the most luminal part of glycocalyx that does allow cell penetration. Increased PBR is considered an accurate index of reduced endothelial glycocalyx thickness because of a deeper RBC penetration in the glycocalyx.
7. Fetuin serum levels, markers of oxidative stress such as malondialdehyde (MDA) serum levels, protein carbonyls aw well as thrombosis and inflammation biomarkers

ELIGIBILITY:
Inclusion Criteria:

* patients with psoriasis
* Age and sex matched patients with CAD, with untreated hypertension and healthy subjects

Exclusion Criteria:

* for psoriasis patients were presence of wall motion abnormalities and ejection fraction ≤ 50%, psoriatic arthritis, history of acute coronary syndrome, familial hyperlipidemia, insulin dependent-diabetes mellitus, chronic obstructive pulmonary disease or asthma, moderate or severe valvular heart disease, primary cardiomyopathies and malignant tumors. CAD was excluded in psoriasis patients by absence of clinical history, angina and reversible myocardial ischemia, as assessed by dobutamine stress echocardiography or thallium scintigraphy
* regarding the group of CAD patients, we only included patients without history of ST elevation myocardial infarction in order to exclude the presence of transmural scar compromising myocardial function indices. Thus, CAD patients with wall motion abnormalities and ejection fraction of ≤ 50% were excluded. In addition, exclusion criteria, were history of acute coronary syndrome without ST-segment elevation within the last year, familial hyperlipidemia, insulin dependent-diabetes mellitus, chronic obstructive pulmonary disease or asthma, moderate or severe valvular heart disease, primary cardiomyopathies and malignant tumor
* in normal controls, CAD was excluded by the presence of normal ECG, absence of clinical history and absence of reversible ischemia by means of treadmill test or dobutamine stress echocardiography

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2014-05-30 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Comparison of effect (improvement or deterioration) of treatment with biological vs. non biological agents on endothelial function in psoriasis | 12 weeks
  Comparison of effect (improvement or deterioration) of treatment with biological agents (anti-tumor necrosis factor-a, anti-interleukin 12/23, anti-interleukin 17A, or apremilast regimen) with the effects of cyclosporine on endothelial function as assessed by flow mediated dilatation of the brachial artery, coronary flow reserve and endothelial glycocalyx thickness
Comparison of effect (improvement or deterioration) of treatment with biological vs. non biological agents on vascular function in psoriasis | 12 weeks
  Comparison of effect (improvement or deterioration) of treatment with biological agents (anti-tumor necrosis factor-a, anti-interleukin 12/23, anti-interleukin 17A, or apremilast regimen) with the effects of cyclosporine on vascular function as assessed by pulse wave velocity, augmentation index and central aortic blood pressure,
Comparison of effect (improvement or deterioration) of treatment with biological vs. non biological agents on cardiac function in psoriasis | 12 weeks
  Comparison of effect (improvement or deterioration) of treatment with biological agents (anti-tumor necrosis factor-a, anti-interleukin 12/23 ,anti-interleukin 17A, or apremilast regimen) with the effects of cyclosporine on cardiac function as assessed by longitudinal myocardial deformation, twisting and untwisting of the left ventricle

SECONDARY OUTCOMES:
Differences and similarities in endothelial function between psoriasis and control groups | 0 and 12 weeks
  Differences in endothelial function between psoriasis and normal controls, and similarities in endothelial function between psoriasis and coronary artery disease patients and untreated hypertension patients before and after 4 week of anti-inflammatory treatment in patients with psoriasis .The following parameters will be compared among the study subgroups endothelial function as assessed by flow mediated dilatation of the brachial artery, coronary flow reserve and endothelial glycocalyx thickness
Differences and similarities in vascular function between psoriasis and control groups | 0 and 12 weeks
  Differences in vascular function between psoriasis and normal controls, and similarities in vascular function between psoriasis and coronary artery disease patients and untreated hypertension patients before and after 4 week of anti-inflammatory treatment in patients with psoriasis .The following parameters will be compared among the study subgroups vascular function as assessed by pulse wave velocity, augmentation index and central aortic blood pressure,
Differences and similarities in cardiac function between psoriasis and control groups | 0 and 12 weeks
  Differences in cardiac function between psoriasis and normal controls, and similarities in cardiac function between psoriasis and coronary artery disease patients and untreated hypertension patients before and after 4 week of anti-inflammatory treatment in patients with psoriasis The following parameters will be compared among the study subgroups cardiac function as assessed by longitudinal myocardial deformation, twisting and untwisting of the left ventricle
Effects of anti-inflammatory treatment on prognosis for major adverse cardiovascular events | 4-year follow-up
  Effects of anti-inflammatory treatment on myocardial infarction, stroke, hospitalization because of heart failure, and cardiovascular death

CONTACTS AND LOCATIONS:
Overall Officials: Ignatios Ikonomidis, Dr, Principal Investigator — University of Athens
Locations (1):
- Attikon Hospital, Athens, Greece

REFERENCES:
- [Derived] Ikonomidis I, Pavlidis G, Lambadiari V, Rafouli-Stergiou P, Makavos G, Thymis J, Kostelli G, Varoudi M, Katogiannis K, Theodoropoulos K, Katsimbri P, Parissis J, Papadavid E. Endothelial glycocalyx and microvascular perfusion are associated with carotid intima-media thickness and impaired myocardial deformation in psoriatic disease. J Hum Hypertens. 2022 Dec;36(12):1113-1120. doi: 10.1038/s41371-021-00640-2. Epub 2021 Nov 25. PMID 34819613
- [Derived] Ikonomidis I, Papadavid E, Makavos G, Andreadou I, Varoudi M, Gravanis K, Theodoropoulos K, Pavlidis G, Triantafyllidi H, Moutsatsou P, Panagiotou C, Parissis J, Iliodromitis E, Lekakis J, Rigopoulos D. Lowering Interleukin-12 Activity Improves Myocardial and Vascular Function Compared With Tumor Necrosis Factor-a Antagonism or Cyclosporine in Psoriasis. Circ Cardiovasc Imaging. 2017 Sep;10(9):e006283. doi: 10.1161/CIRCIMAGING.117.006283. PMID 28899951